CLINICAL TRIAL: NCT01326845
Title: A Multicenter, Randomized, Comparative Study of Different Deferasirox Administration Regimens on Gastrointestinal (GI) Tolerability in Low or Intermediate (Int-1) Risk MDS Myelodysplastic Syndrome Patients With Transfusional Iron Overload.
Brief Title: Myelodysplastic Syndrome (MDS) Gastrointestinal (GI) Tolerability Study
Acronym: MACS1574
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated due to insufficient enrollment.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2417; 2011-001077-13 (EudraCT Number)
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Myelodysplastic Syndrome; Transfusional Iron Overload
Keywords: Gastrointestinal adverse events,; myelodysplastic syndrome,; transfusional iron overload diarrhea,; constipation abdominal pain,; vomiting
MeSH Terms: conditions — Myelodysplastic Syndromes; Vomiting | interventions — Deferasirox

ARMS (2):
- Deferasirox am (Experimental): Deferasirox 20 mg/kg/day taken in the morning, 30 minutes before food
  Interventions: Drug: Deferasirox
- Deferasirox pm (Experimental): Deferasirox 20 mg/kg/day taken in the evening, no less than 2 hours after the last food intake or at least 30 minutes before the evening meal
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox
  Other Names: ICL670

SUMMARY:
The objective of the study is to evaluate and compare the frequency and severity of GI adverse events in different dose administration regimens. The patient population consists of low or intermediate (int-1) risk myelodysplastic syndrome (MDS) patients with transfusional iron overload. The study patients are randomized to either a morning dose of 20 mg/kg/day deferasirox or an evening dose of the same. Patients are then followed up for 6 months for any GI events and are assessed using patient reported outcomes tools e.g. a patient diary.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any screening procedures
* Male or female patients ≥ 18 years of age
* Patient must weigh between 45-135 kg
* Patients with low or intermediate (int-1) risk MDS, as determined by IPSS score or RA, RARS by WHO criteria. IPSS must be confirmed by a bone marrow examination within 6 months prior to study entry and must be hematologically stable

Deferasirox naïve:

Sexually active pre-menopausal female patients must use double-barrier contraception, oral contraceptive plus barrier contraceptive, or must have undergone clinically documented total hysterectomy and/or oophorectomy, tubal ligation

Exclusion Criteria:

* History or current GI disease
* Systemic diseases which could prevent study treatments
* Left ventricular ejection fraction< 50 % by echo cardiography
* Serum creatinine > 1.2 x ULN at screening
* Platelet counts < 25x 109/L except in cases where guidance is already given in the local deferasirox label
* AST or ALT > 2.5 xULN at screening

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- France (5):
  - Novartis Investigative Site, Caen, Cedex
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Italy (3):
  - Novartis Investigative Site, Alessandria, AL
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Roma
- Novartis Investigative Site, Bloemfontein, South Africa
- Novartis Investigative Site, Madrid, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deferasirox am | Deferasirox pm
Started | 7 | 5
Completed | 0 (Study terminated early) | 0 (Study terminated early)
Not Completed | 7 | 5
Not completed — Administrative Problems | 5 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Misisng | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferasirox am | Deferasirox pm | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (7.5) | 71.6 (8.65) | 70.5 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Frequency of Overall Newly Occurring GI Adverse Events (AEs) in the Two Treatment Arms
Description: Study was prematurely terminated and not powered for efficacy. Frequency of GI AEs during the overall study period is available in the AE tables reported in the safety section.
Time Frame: 3 months
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Difference in Frequency of Overall Newly Occurring GI AEs Between the Two Treatment Groups at Month 6.
Description: Study was prematurely terminated and not powered for efficacy.
Time Frame: 6 months
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Difference in Frequency of Specific Commonly Reported GI AEs Between the Two Treatment Groups
Description: Study was prematurely terminated and not powered for efficacy.
Time Frame: months 3 and 6.
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Difference in Severity of Overall GI AEs Between the Two Treatment Groups
Description: Study was prematurely terminated and not powered for efficacy.
Time Frame: months 3 and 6.
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Difference in Severity of Specific Commonly Reported GI Symptoms Between the Two Treatment Groups
Description: Study was prematurely terminated and not powered for efficacy.
Time Frame: months 3 and 6
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Difference in Frequency and Severity of All Non-GI AEs Between the Two Treatment Groups
Description: Study was prematurely terminated and not powered for efficacy.
Time Frame: months 3 and 6
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: the Difference Between the Time From Baseline to the First Occurrence of GI AEs Between the Two Treatment Groups
Description: Study was prematurely terminated and not powered for efficacy.
Time Frame: 3 months, 6 months
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Difference in Severity of GI Symptoms, Bowel Habits and Level of Satisfaction From the Patient's Perspective Between the Two Treatment Groups
Time Frame: 3 months, 6 months
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Difference in Reducing Serum Ferritin After Each Month of Study Drug Administration Between the Two Groups
Description: Study was prematurely terminated and not powered for efficacy.
Time Frame: 3 months, 6 months
Arm/Group | Deferasirox am | Deferasirox pm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- ICL am: ICL am
- ICL pm: ICL pm
Arm/Group | ICL am | ICL pm
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/5
Other Adverse Events (participants affected / at risk) | 5/7 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICL am (N=7) | ICL pm (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ICL am (N=7) | ICL pm (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 2 | 0
Lyme disease (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.